CLINICAL TRIAL: NCT06831669
Title: Metabolomic Profiles as Predictors of Treatment Response and Toxicities in Locally Advanced Rectal Cancer Undergoing Total Neoadjuvant Therapy
Brief Title: Metabolomics to Predict Treatment Response and Toxicities in Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG3P0091
Record Dates: First submitted 2024-01-16; First posted 2025-02-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Rectal Neoplasm Malignant
Keywords: Rectal cancer; Total neoadjuvant therapy; Metabolomics; Radiation proctitis
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood, urine, faecal, and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Collecting biospecimens — Collecting blood, urine, tissue, and faecal samples

SUMMARY:
Background: Colorectal cancer is the leading cause of cancer-related deaths in Taiwan, with rectal cancer accounting for approximately 27% of all cases. Total neoadjuvant therapy (TNT), which consists of chemotherapy and radiation therapy delivered before surgery, has become the standard of care for locally advanced rectal cancer. However, there is currently no reliable method for predicting the response to TNT or the occurrence of radiation proctitis, a common side effect of treatment.

Objective: This study aims to evaluate the metabolomic profiles of individuals with locally advanced rectal cancer undergoing TNT and to identify a panel of metabolites that can predict treatment response and toxicities.

Methods: A prospective cohort study will be conducted to enrol patients with locally advanced rectal cancer who are scheduled to receive TNT. Blood, urine, tissue, and faecal samples will be collected at baseline, during, and after chemoradiotherapy. Metabolomic profiling of the samples will be performed using liquid-chromatography mass spectrometry (LC-MS). Treatment response will be assessed based on clinical downstaging (defined as a decrease in tumour size and/or T and N stage after TNT) and pathological response, such as pathological complete response (pCR). Radiation proctitis will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. PCA and PLSDA will be used to identify metabolites that are associated with treatment response and radiation proctitis. Receiver operating characteristic (ROC) curves will be used to assess the predictive performance of the identified metabolites. Univariate and multivariate logistic regression will be used to build models to predict treatment response and radiation proctitis.

DETAILED DESCRIPTION:
Hypothesis: Metabolomic profiling can be used to predict the response to total neoadjuvant therapy (TNT) and the incidence of radiotherapy-related diarrhoea in patients with locally advanced rectal cancer.

Rationale of the project: Metabolomics is a powerful tool for identifying biomarkers that are associated with disease and treatment response. It is more closely related to the biological phenotype than other omics approaches, such as genomics and transcriptomics, and it has the potential to be used for precision health applications.

In this project, the investigators aim to use metabolomics to predict the response to total neoadjuvant therapy (TNT) and the incidence of treatment-related toxicity in rectal cancer patients prior to treatment. This would allow us to select patients who are most likely to benefit from TNT and to minimize the risk of complications.

There is a growing body of evidence that suggests that metabolomics can be used to predict treatment response and toxicity in cancer patients. For example, one study found that plasma metabolites could be used to predict the overall survival and progression-free survival of patients with colorectal cancer. Another study found that the level of pretreatment faecal butyrate was directly related to gastrointestinal toxicity in prostate cancer patients. However, most studies on metabolomics and cancer have used long-course chemoradiotherapy. There is a limited amount of research on the use of metabolomics to predict treatment response and toxicity to TNT.

This project is the first to comprehensively evaluate the metabolomic profiles of patients with locally advanced rectal cancer undergoing TNT at multiple time points during and after treatment using liquid chromatography-mass spectrometry (LC-MS), and to assess the association of these profiles with treatment response and toxicities. The findings from this study have the potential to lead to the development of non-invasive biomarkers for predicting treatment response and toxicities, which could improve the clinical management of rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum
* Scheduled to receive total neoadjuvant therapy

Exclusion Criteria:

* Previous pelvic radiation therapy
* Inflammatory bowel disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will prospectively recruit 250 patients with locally advanced rectal cancer who are scheduled to receive total neoadjuvant therapy (TNT) at Chang Gung Memorial Hospital, Linkou, over a two-year period from 2024 to 2025. Blood, urine, fecal, and tissue samples will be collected from patients at baseline, during, and after TNT.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2028-12-12 (Estimated); Study Completion 2033-12-12 (Estimated)

PRIMARY OUTCOMES:
Predictive Accuracy of Metabolomic Profiles for Complete Response (CR) | From enrollment to surgical resection or up to 6 months after completion of radiotherapy (whichever occurs first)
  Sensitivity, specificity, positive predictive value, negative predictive value, and overall accuracy of metabolomic signatures in predicting complete response (CR). For patients undergoing surgical resection, CR will be determined based on histopathological examination of resected specimens (pathological CR). For patients who do not undergo surgery, clinical CR will be defined by findings from digital rectal examination (DRE), colonoscopy, and imaging studies (e.g., MRI or CT) up to six months after radiotherapy completion.

SECONDARY OUTCOMES:
Number of Participants With Grade 3-4 Treatment-Related Toxicities as Assessed by CTCAE | From initiation of radiotherapy to 21 days after completion.
  Incidence of severe (Grade 3-4) toxicities associated with radiotherapy, as determined by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE version 5.0).

OTHER OUTCOMES:
Changes in Metabolomic Profiles From Baseline to Post-Radiotherapy | At baseline, and within two weeks and three months following completion of radiotherapy.
  Alterations in identified metabolomic biomarkers (e.g., normalised intensities of specific metabolites measured by LC-MS) between baseline and post-radiotherapy time points. Reported as changes in metabolite intensities (e.g., mean, median, or fold change) compared to baseline measurements.
Correlation Between Changes in Metabolomic Biomarkers and Grade 3-4 Toxicities | From baseline to 21 days after completion of radiotherapy.
  Correlation (e.g., Pearson's or Spearman's correlation coefficient) between alterations in metabolomic profiles and the incidence of Grade 3-4 toxicities during and immediately following radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan